CLINICAL TRIAL: NCT02675634
Title: Investigation of Two New 1-piece Ostomy Products in People With an Ileostomy or Colostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP266
Record Dates: First submitted 2016-01-29; First posted 2016-02-05 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Ileostomy; Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Test A, Test B, Subjects own product (Experimental): The subjects first test Coloplast Test A, followed by Coloplast Test B and finally Subjects own product
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Subjects own product
- Test A, Subjects own product, Test B (Experimental): The subjects first test Coloplast Test A, followed by Subjects own product, and finally Coloplast Test B
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Subjects own product
- Test B, Test A, Subjects own product (Experimental): The subjects first test Coloplast Test B, followed by Coloplast Test A and finally Subjects own product
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Subjects own product
- Test B, Subjects own product, Test A (Experimental): The subjects first test Coloplast Test B, followed by Subjects own product, and finally Coloplast Test A
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Subjects own product
- Subjects own product, Test A, Test B (Experimental): The subjects first test Subjects own product, followed by Test A, and finally Coloplast Test B
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Subjects own product
- Subjects own product, Test B, Test A (Experimental): The subjects first test Subjects own product, followed by Test B, and finally Coloplast Test A
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Subjects own product

INTERVENTIONS:
Device: Coloplast Test A — Test A is a new 1-piece ostomy appliance developed by Coloplast A/S
Device: Coloplast Test B — Test B is a new 1-piece ostomy appliance developed by Coloplast A/S
Device: Subjects own product — The comparator product is the ostomy appliance product that the subject normally uses. This could include products like SenSura , SenSura Mio, Confidence Natural, Moderma Flex and many more. data from the subject own product will be pooled so they appear as one comparator group.

SUMMARY:
This clinical investigation is intended to explore the performance and safety of two newly developed ostomy products with regard to the products fit to body properties.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and in DK: signed a letter of authority 2. Are at least 18 years of age and have full legal capacity 3. Have had their ileostomy or colostomy for at least 3 months 4. Are able to use a baseplate cut-max 15 to 40 mm 5. Are able to handle the product themselves 6. Currently using a 1-piece flat product 8. Willing to use an open bag size maxi during the investigation 9. Are able to use a custom cut (custom fit) product 10. Are suitable for participating in the investigation - this means that the subjects must be able to follow all elements of the study procedures.

Exclusion Criteria:

1. Are currently receiving or have within the past 2 months received radio-and/or chemotherapy (low doses chemotherapy are allowed for other indications than cancer, e.g. below 15 mg methotrexate for rheumatoid arthritis)
2. Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area, e.g. lotion or spray. Systemic steroid treatment (e.g. injection, or tablet) are allowed.
3. Are pregnant or breastfeeding**
4. Are participating in other interventional clinical investigations or have previously participated in this investigation
5. Use irrigation during the investigation (flush the intestines with water, this is mostly for people with a colostomy)
6. Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)
7. Have a loop ostomy (also called double barrel ostomy)
8. Have known hypersensitivity towards any of the products used in the investigation

   * In DK: women in the child-bearing age will be ask to produce a negative pregnancy test and to sign a form ensuring the use of safe contraception during the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla F Vibjerg, Study Chair — Head of Clinical Operation
Locations (12):
- United States (3):
  - Radiant Research, Tempe, Arizona
  - Prism research center, Saint Paul, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
- TFS, Søborg, Denmark
- QPS Netherlands, Groningen, Netherlands
- United Kingdom (7):
  - Synexus Midlands, Birmingham
  - Pilgrim Hospital, Boston
  - Illingworth Research Nurses, Cheshire
  - Lincon Country hospital, Lincoln
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Kettering General hospital, Northamptonshire
  - Synexus Hexam, Northumberland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited through the Coloplast A/S database and from hospital sites
Period: Test Period 1
Arm/Group | Test A, Test B, Subjects Own Product | Test A, Subjects Own Product, Test B | Test B, Test A, Subjects Own Product | Test B, Subjects Own Product, Test A | Subjects Own Product, Test A, Test B | Subjects Own Product, Test B, Test A
Started | 10 | 8 | 9 | 9 | 10 | 9
Completed | 10 | 7 | 8 | 8 | 10 | 9
Not Completed | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Device deficiency that did not lead to A | 0 | 0 | 1 | 0 | 0 | 0
Period: Test Period 2
Arm/Group | Test A, Test B, Subjects Own Product | Test A, Subjects Own Product, Test B | Test B, Test A, Subjects Own Product | Test B, Subjects Own Product, Test A | Subjects Own Product, Test A, Test B | Subjects Own Product, Test B, Test A
Started | 10 | 7 | 8 | 8 | 10 | 9
Completed | 9 | 7 | 8 | 8 | 10 | 8
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Test Period 3
Arm/Group | Test A, Test B, Subjects Own Product | Test A, Subjects Own Product, Test B | Test B, Test A, Subjects Own Product | Test B, Subjects Own Product, Test A | Subjects Own Product, Test A, Test B | Subjects Own Product, Test B, Test A
Started | 9 | 7 | 8 | 8 | 10 | 8
Completed | 9 | 7 | 8 | 8 | 10 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consist of all enrolled subjects
Groups:
- The Study Population: This consists of all participants who were enrolled in the study
Arm/Group | The Study Population
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject did not aswer the gender question therefore this information is missing.
  Participants
    number analyzed (Participants) | 54
    Female | 14
    Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Fit to Body
Description: Subjects will evaluate the fit to body for each product by answering the question "how was the baseplates ability to fit the body contours in the area around the stoma?" The question is answered using an ordinal 5 point scale ranging from very poor to very good. The result shown below shows the fraction of subject who answered 'Good' or' Very Good' to the question.
Time Frame: 14 +/- 2 days
Measure: Number; unit: percentage of good or very good
Groups:
- Test A: This is the result from all subjects evaluating Test A
- Test B: This is the results from all the subjects evaluating Test B
- Own Product: this is the result from all the subjects evaluating Own product.
Arm/Group | Test A | Test B | Own Product
Number analyzed (Participants) | 51 | 54 | 51
percentage of good or very good | 93 | 88 | 57

ADVERSE EVENTS:
Time Frame: Adverse events were collected from subject enrollment to the subject left the study. Subjects with serious adverse events were followed until their condition was resolved.
Arm/Group | Test A | Test B | Own Product
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 8/52 | 11/54 | 4/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A (N=52) | Test B (N=54) | Own Product (N=51)
Obstibation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A (N=52) | Test B (N=54) | Own Product (N=51)
Peristomal skin dermatitis (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (12) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less